

Statistical Analysis Plan

NCT Number: NCT05932407

Title: A Cohort Study to Compare the Risk of Hemorrhage (Serious Intracranial Hemorrhage Such as Cerebral Hemorrhage and Subarachnoid Hemorrhage) Between Trintellix Tablets and SSRIs in Patients With Depression Using JMDC Claims Database

Study Number: Vortioxetine-4005

Document Version and Date: Version 2.0 / 28-Aug-2024

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

Note; This document was translated into English as the language on original version was Japanese.

# statistical analysis plan

Patients with depression using the medical information database, JMDC claims database and patients with depression

A Cohort Study to Compare the Risk of Haemorrhage (Serious Intracranial Haemorrhage Such as Cerebral Haemorrhage and Subarachnoid Haemorrhage) between Trintellix Tablets, SSRI and in only and subject to

Vortioxetine-4005

Takeda Pharmaceutical Company Limited.

| Preparation | Date of signature | Signature |
|-------------|--------------------------|-----------|
| | 28-8-2024 15:59:21 JST | |
| Approval | Date of signature | |
| прргоча | | |
| | 28-8-2024 16:40:17 JST | |

| . Preparation | /Dovicion | Docord |
|---------------|------------|--------|
| . Preparadon | / Revision | Record |

| Version | Key Changes | Reason for change | |
|---|---|---|---|
| [VERSION DATE] | | | |
| 1.0 | New document | • | 150 |
| [2024/3/25] | | | 15 |
| L - /-/ -1 | | | $\mathcal{O}_{\mathcal{O}}$ |
| | | | 0) |
| 2.0 | 6.5 Sensitivity analysis 2) | Based on the agreements from the PMDA consultation (PMDA | S |
| page 48), sensitivit | y [2024/8/28] was determined. | The conditions for analysis were changed as follows. Changes are | in |
| underlined. | | | SI |
| | | < Before change > | |
| | | 2) GRACE PERIOD CHANGE | |
| | | After changing Grace Period to up to 90 days, the analysis set (analysis s | et |

Property of Takeda. For non-commercial use

After changing Grace Period to up to 90 days, the analysis set (analysis set [sensitivity analysis 2)) will be reorganized, and the same analyses as the case performed.

< After change >

Change Gap Period and Graee Period to "Up to 90 Days."

and changed to the analysis population (analysis population)

(Sensitivity analysis, 2) and will be reorganized, and the same analyses as the Case composition diagram, patient background, and primary analysis will be performed.

Summary of the survey and summary of the statistical analysis plan

| Product name | TRINTELLIX Tablets 10 mg, 20 mg | |
|---|---|---|
| Survey title | Haemorrhages associated with TRINTELLIX Tablets and SSRIs in patients with depression using the medical information database JMDC claims database (serious headache including cerebral haemorrhage and subarachnoid haemorrhage) | |
| | Cohort study to compare the risk of intradermal bleeding | |
| Type of investigation | Post-marketing database survey | |
| Purpose of inspection | To evaluate the relative risk of serious intracranial hemorrhage requiring hospitalization in patients with depression treated with TRINTELLIX Tablets compared to SSRI in approximately 3 years from the launch date of TRINTELLIX Tablets (November 2019 to November 2022). | reims of U |
| Medical information data used for<br>survey <i>Tano</i> t '— | JMDC Claims Database will be used. This database has receipt data and health checkup data provided by multiple health insurance societies. The cumulative population is approximately 14 million (as of May 2022). | ) |
| Survey period (data period) | Data period: November 1, 2018 to November 30, 2023 Enrollment period: November 27, 2019 to November 30, 2022 | |
| Study design | Cohort design | |
| Scope of patients to be surveyed | Patients with depression | |
| Definitions of Exposure and Control<br>Groups | Among the subjects selected according to the inclusion/exclusion criteria, the group of patients who were prescribed TRINTELLIX Tablets on the first day of prescription is defined as the exposure group, and the group of patients who were prescribed SSRI is defined as the control group. | |
| Outcome | Regarding serious intracranial hemorrhage requiring hospitalization, there are 3 definitions combining injury/disease code (ICD-10 code), therapeutic drug (drug code based on medical service fee points), and medical practice (Hospitalization record, classification code). | |
| | For the primary analysis, incidence rates (per 10,000 person-years) of the outcome during the follow-up period will be estimated in the exposure and control groups, and hazard ratios (crude and adjusted) with reference to the control group will be calculated using Cox proportional hazards models. The following analyses will be performed for secondary analyses: Kaplan-Meier Time to Outcome Measures | |
| Lakeda. For non | <ul> <li>Estimated Incidence Rates (/ 10,000 PY) of Outcomes by SSRI Components in the Control Group</li> <li>Analysis similar to the primary analysis with alternative definition of outcome</li> <li>The following analyses will be performed as sensitivity analyses:</li> <li>Look back period. Analysis similar to the primary analysis with different definitions of gap period, grace period, and outcome</li> </ul> | |
| | <ul> <li>The propensity score for each patient will be estimated using a logistic regression model with cohort as an objective variable and all covariates as explanatory variables, and the hazard ratio relative to the control group will be calculated using a Cox proportional hazards model with cohort and propensity score as two variables in the model.</li> </ul> | |

### TABLE OF CONTENTS

| List o | f Abb | previations | 6 |
|---|---|---|---|
| Defin | itions | s of Terms | 6 |
| <b>1.</b> 1 | Purpo | ose and Scope | 7 |
| | • | • | 50 |
| | amp | ole Size and Rationale | |
| 3. 9 | Study | population | 7 |
| <b>4.</b> 1 | Defin | ition of analysis sets and variables | 8 CETHES |
| 4. | 1. | Study Population Definitions | 8 |
| | 4.1. | .1. Period covered | 8 |
| | 4.1. | .2. Population Entry Criteria | 8 |
| | 4.1. | 3. Population Exclusion Criteria | 8 |
| 4. | 2. | Study Population Definitions | 8 |
| | 4.2. | .1. Exposure | 8 |
| | 4.2. | | 8 |
| 4. | 3. | Observation period | 8 |
| | 4.3. | 1. Duration of prescription | 8 |
| | 4.3. | 2 Start date and end date of observation period | q |
| | 4.3. | .3. Follow-up period | 9 |
| 4. | 4. | 3. Follow-up period | 9 |
| 4. | <b>7</b> | Lovariates | 11 |
| | | Descriptive statistics | 40 |
| 5. ( | jENE | RAL STUDY CONSIDERATIONS | 13 |
| 5. | 1. | Descriptive statistics | 13 |
| 5. | 2. | Display of numerical values | 13 |
| 5. | 3. | Software Used for Aggregate Analysis | 13 |
| 5. | 4. | Significance level and confidence interval | 13 |
| 5. | 5. | Handling of missing data | 13 |
| 5. | 6. | Handling of Outliers | 13 |
| <b>6</b> . <i>1</i> | Analy | vsis Methods | |
| 6. | 1 | Patient composition | 1.4 |
| 6. | | Patient characteristics | |
| 6. | | Primary Analysis | |
| 6. | | | |
| 6. | | Secondary Analyses Sensitivity analyses | |
| ο. | J. 6 | Sensitivity analyses | 15 |
| 7, 4 | <b>YPPE</b> | NDICES | 17 |
| 7. | 1. | References | 17 |

Property of Takeda: For non-commercial use only and subject to the applicable Terms of Use

## List of Abbreviations

| Abbreviation | Official name | Japanese name |
|---|---|---|
| SSRI | Selective Serotonin Reuptake Inhibitor | selective serotonin reuptake inhibitor |
| NSAID | Non-Steroidal Anti-Inflammatory Drug | Non-Steroidal Anti-Inflammatory Drugs |
| DB | Database | Database |
| ICD | | International Statistical Classification of Diseases and Related Health<br>Problems |
| СТ | Computed Tomography | computed tomography |
| MRI | Magnetic Resonance Imagin | magnetic resonance imaging |
| MRA | Magnetic Resonance Angiography | magnetic resonance angiography |

## **Definitions of Terms**

| MRA | Magnetic Re | sonance Angiography | magnetic resonance angiography |
|---|---|---|---|
| | | | The app. |
| Defin | itions of Te | erms | *O |
| Т | l'erm | | Definition |
| Index date | | Date of first prescription within enrollment period | (b) |
| Look back period | I | Period of Measurement of Each Covariate, etc. | 450 |
| Observation pe | | Period during which each subject will be observed (look bath Period from the date of each prescription to the date of comprescription -1) | ck period+ follow-up period)<br>npletion of prescription (date of prescription + number of days of |
| Duration of pro | escription | How long the prescription is considered to be ongoing | |
| Gap Period | | The period between consecutive prescribed periods | |
| Grace Period | | Additional period to be added as the prescription continual missed doses and persistent effects of discontinued drugs | tion period after the end of the prescription period in consideration of |
| Follow-up peri | iod | Period during which each subject will be followed up to con<br>after the Index Date to the day of completing the observation | nfirm the presence or absence of occurrence of outcomes (from the day on period) |
| Data period | | Period during which target data for this survey are extracted | ed from the database |
| Launch Date | | This drug launched on November 27, 2019 | |
| This DB MDC Claims Database | | | |
| This drug TRINTELLIX Tablets 10 mg and TRINTELLIX Tablets 20 mg | | | |
| Health insuran | ice claims | Medical hospitalization receipt or DPC receipt (inpatient), (dispensing) | nedical non-hospitalization receipt (outpatient), dispensing receipt |

### 1. Purpose and Scope

This study will evaluate the relative risk of this drug serious intracranial hemorrhage requiring hospitalization during 3 years from the launch date of this drug (2019, November, until 2022, and November) in patients with depression compared with during SSRI treatment.

### 2. Sample Size and Rationale

As a result of the feasibility survey conducted using this DB prior to this survey, \* the number of patients with depression requiring medication in 2019, November (launch date), - 2022 and January was approximately 172,000, and the number of patients in the exposure and control groups to whom the inclusion/exclusion criteria were applied was approximately 11,000 and 76,000, respectively. Considering that the enrollment period in this survey will be up to 2022 or November, approximately 14,000 and 101,000 subjects are expected to be enrolled in this drug and control groups, respectively.

According to a report by Renoux et al., using the Clinical Practice Research Datalink in the UK, over 1.36 million adults who first started taking an SSRI or tricyclic antidepressant between January 1 and June 30, 2014 1995 were followed up for an average of 5.8 years. During the follow-up period, 3,036 patients were diagnosed with intracranial hemorrhage (3.8 cases per 10,000 people per year, or an incidence rate of 0.00038 per 1 year), and it was reported that the risk of intracranial hemorrhage in SSR1 was increased by 17% compared to tricyclic antidepressants 1]. Since the incidence of cerebral haemorrhage is 2.4 times higher in Asians than in non-Asians, the incidence of intracranial haemorrhage per 1 year in SSRI estimated in the Japanese survey was assumed to be 0.0009.

In contrast, using the sample size calculation formula 6.9 proposed for comparative studies in post-marketing surveillance in Sample Size Design for Medicine, a sample size of 13,242 exposed (this drug) and 92,694 unexposed (control) patients can be calculated to detect a 2 -fold increase in the rate of intracranial hemorrhage with TRINTELLIX compared to an SSRI (i.e., a further 0.0009 increase in the rate per 1 year of intracranial hemorrhage), assuming a randomization ratio of 7: 1 for the control group versus this drug group, a two-sided significance level of (4) 0.05, and a power of (1-8) 0.8 (When the one-sided significance level was 0.05, the sample sizes were 10,644 and 74,508 subjects, respectively.).

Thus, taking into account the accumulation of data, etc. in the future, it is considered that this study can be sufficiently conducted using this study, DB, and MT-MD001.

\*1: Protocol Appendix 4 Information on the number of patients, etc. subject to the survey that can be obtained from the medical information database

(that) and 2)

### Study population

Patients with depression registered in JMDC Claims Database

### 4. Definition of analysis sets and variables

### 4.1. Study Population Definitions

### 1.1 .1. Period covered

Data period: November 1, 2018 to November 30, 2023

Enrollment period: November 27, 2019 (date of launch) to November 30, 2022

### 4.12 Population Entry Criteria

Patients must meet all of the following criteria to be eligible for enrollment in the study:

- 1) Diagnosed with depression and prescribed this drug or SSRI during the enrollment period (Index date: Date of first prescription during enrollment period).
  - 2) It is possible to observe the (180 days) or (look back period) for the past 6 months from the day before the Index date.
  - 3) No this drug or SSRI or was prescribed during the look back period.

### 4.13 Population Exclusion Criteria

Patients meeting any of the following criteria will be excluded.

1) Look back period Intracranial hemorrhage was diagnosed.

See "4.4. Outcome Definition (Definition 2)" for the diagnosis of intracranial hemorrhage.

- 2) Index date, this drug, SSRI, and are used concomitantly.
- 4.2. Study Population Definitions

### 4.2.1. Exposure

Of patients in the target population, patients for whom this drug was prescribed on the Index date and patients

### 4.2.2. Control group

Patients in the target population who are given a prescription of SSRI on the Index date

### 4.3. Observation period

### 4.3.1. Duration of prescription

Prescription continuation period is the period from the day after the Index Date to (Grace Period) after 30 days from the final prescription completion date. In addition,

If the interval (Gap Period) between consecutive prescription periods is within 30 days, the prescription is considered to be continued. If the interval (Gap Period) between consecutive prescription periods is 31 days or more, the prescription is considered to be discontinued.

### **4.3.2.** Start date and end date of observation period

First day of observation period: The day before 6 months in the past (180 days) from the day before Index Date

End date of observation period: among the following, Index date, the earliest date after

- (1) Onset of outcome (intracranial hemorrhage)
- (2) End of prescription period for this drug or SSRI End of prescription period for
- (3) Switching to other drugs (this drug or), SSRI, and switching to
- (4)With this drug, SSRI and combination
- (5) Death
- (6)Withdrawal from health insurance society or termination of the agreement between health insurance society and the stock company, JMDC and JMDC
- 7 From the day after Index Date to Day 360 (end of follow-up period)

### 4.3.3. Follow-up period

First day of the follow-up period: Index date the day after

End date of follow-up period: End date of observation period

Follow-up period: the end date of follow-up period - the start date of follow-up period + 1

### 4.4. Outcome definitions

Outcome is defined as intracranial haemorrhage such as serious cerebral haemorrhage and subarachnoid haemorrhage requiring inpatient treatment that meets all of the conditions in the following definitions.

Definition 1:

- 1) ICD-10 code: 4) 5) with a record of ICD -10 code for any of 160 subarachnoid hemorrhage, 161 intracerebral hemorrhage, or 162 other nontraumatic intracranial hemorrhage. (excluding those with suspicion flag)
- 2) There is a record of hospitalization ("hospitalization or DPC in" receipt type ") in the same month as the diagnosis of intracranial haemorrhage such as cerebral haemorrhage and subarachnoid haemorrhage in 1) above.
- 3) A record of any of CT, MRI, or MRA tests (Category code: E 200, computed tomography (CT) imaging (per series), E 202, magnetic resonance computed tomography (MRI) imaging (per series), E 203, computed tomography) is present within the same hospitalization (the same "Receipt ID) for intracranial haemorrhage such as cerebral haemorrhage and subarachnoid haemorrhage mentioned in 2) above.

(date of outcome onset)

### Definition 2:

- In addition to the above definition for Definition 1, any of the following records (1) to (6) is present within the same hospitalization (the same receipt) for intracranial hemorrhage such as cerebral hemorrhage and subarachnoid hemorrhage according to Definition 12).
- (1)Anti-edema agents: Drug Code K01F1 (for osmotherapy) 6)

- clazosentan sodium (C04A1)].
- craniectomy, K 164 intracranial hematoma evacuation (Craniotomy, K 176 Cerebral aneurysm inflow vessel clipping (Performed through craniotomy, K 178, cerebrovascular procedure)) 5) 6)

Definition 3:

- ICD-10 code: documented ICD -10 code for either intracranial hemorrhage (160 Subarachnoid haemorrhage, 161 Intracerebral haemorrhage 162 Other non-traumatic intracranial haemorrhage) or gastrointestinal hemorrhage (1850 Esophageal varices with hemorrhage, K 226 Esophagogastric junction laceration bleeding syndrome, K 250 Gastric ulcer/acute with hemorrhage, K 251 Gastric ulcer/acute with hemorrhage and perforation, K 252 Gastric ulcer/acute with both hemorrhage and perforation, K 253 Gastric ulcer/acute without hemorrhage or perforation, K 254 Gastric ulcer/chronic or unspecified with hemorrhage, K 255 Gastric ulcer/chronic or unspecified with perforation, K 256 Gastric ulcer/chronic or unspecified with both hemorrhage and perforation, K 260 Duodenal ulcer/acute with hemorrhage, K 261 Duodenal ulcer/acute with perforation, K 262 Duodenal ulcer/acute with both hemorrhage and perforation, K 250 Duodenal ulcer/acute, without hemorrhage or perforation, K 251 Duodenal ulcer/chronic or unspecified, with hemorrhage, K 252 Duodenal ulcer/chronic or unspecified, with perforation, K 253 Duodenal ulcer/chronic or unspecified, with both hemorrhage and perforation, K 254 Peptic ulcer of unspecified site/acute, with hemorrhage, K 255 Gastrojejunal ulcer/chronic or unspecified, with hemorrhage, K 256 Gastrojejunal ulcer/chronic or unspecified, with perforation, K 260 Acute hemorrhagic gastritis, K 1850 Hematemesis, K 226 Melaena, K 263 Gastrointestinal hemorrhage, unspecified). (excluding those with suspicion flag)
- Property of Fakeda. For non-commen 2) There is a record of hospitalization ("hospitalization or DPC in" receipt type) in the same month as the diagnosis of intracranial haemorrhage or gastrointestinal haemorrhage such as cerebral haemorrhage and subarachnoid haemorrhage in 1) above.

### 4.5. Covariates

The following covariates will be used to adjust the background of the exposure and control groups (COV 1 and 2 will be used for multivariate analysis, and COV  $1 \sim 3$  will be used for propensity score analysis.).

| | Table (4) -1 Covariates |
|---|---|
| Covariate Name | Time of adoption/method of derivation |
| COV1 | · C |
| Age (continuous variable) patient data. | Age as of the Index Date is calculated from the month and year of birth of the Participant in the |
| Gender (Male, Female) | Obtained from the sex of subscribers in patient data |
| COV2 | |
| Prescription of administration of antithrombotic drug (Yes, No) | If there is at least 1 relevant prescription information on [Index date-30] to [Index date-1], Yes. None if there is no applicable data. |
| Prescribed NSAID use (Yes, No) | [! ^ Early -30] If there is at least 1 relevant prescription information in 10 [-1 in 1 year], Yes. None if there is no applicable data. |
| Hypertension (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |
| cov3 | enb. |
| Atypical antipsychotic prescription (Yes, No) | If there is at least 1 relevant prescription information on [Index date-30] to [Index date-1], Yes. None if there is no applicable data. |
| Prescription of administration of phenothiazine antipsychotics (Ye date-1], | es, No) If there is at least 1 relevant prescription information on [Index date-30] to [Index Yes, None if there is no applicable data. |
| Tricyclic antidepressant prescription (Yes, No) | If there is at least 1 relevant prescription information on [Index date-30] to [Index date-1], Yes. None if there is no applicable data. |
| Diabetes mellitus (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |
| Ischaemic heart disease (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |
| Ischemic cerebral infarction (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |
| Cerebral amyloid angiopathy (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |
| Cerebral aneurysm (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |
| Brain tumor (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |
| Epilepsy (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |
| Hepatic disease (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. 1 None if there is no applicable data. |

| Renal failure (Yes, No) | Yes, if at least one diagnosis of the disease is available during the look back period. $\boldsymbol{1}$ |
|---|---|
| | None if there is no applicable data. |
| Alcoholism (Yes, No) | Yes, if at least one diagnosis of the disease is available during the look back period. $\boldsymbol{1}$ |
| | None if there is no applicable data. |
| Bleeding from the nose (Yes, No) | Yes, if at least one diagnosis of the disease is available during the look back period. $\boldsymbol{1}$ |
| | None if there is no applicable data. |
| Dyslipidemia (Yes, No) | Yes, if at least one diagnosis of the disease is available during the look back period. 1 |
| | None if there is no applicable data. |
| Obesity (Yes, No) | Yes, if at least one diagnosis of the disease is available during the look back period. 1 |
| | None if there is no applicable data. |
| Metabolic syndrome (Yes, No) | Yes, if at least one diagnosis of the disease is available during the look back period $oldsymbol{1}$ |
| | None if there is no applicable data. |
| Sleep apnoea syndrome (Yes, No) | Yes, if there is at least one diagnosis of the disease in the look back period. $1$ |
| | None if there is no applicable data. |
| Peripheral Arterial Disease (Yes, No) | Yes, if at least one diagnosis of the disease is available during the look back period. 1 |
| | None if there is no applicable data. |
| Drinking history (Present, absent, unknown) | In the health checkup data during the look back period, |
| | <ul> <li>If there is a description of "Drinking alcohol: every day" or Drinking alcohol: at least<br/>1Gou" in at least one case</li> </ul> |
| | Yes, Yes |
| | - "Drink: sometimes 0r, hardly drink" and "Drink amount: less than 1Gou" |
| | None if there is only description |
| | Otherwise, unknown |
| Smoking history (Present, absent, unknown) | In the health checkup data during the lookback period, |
| | Yes if smoking is described in at least one case. |
| | Absent if there is only a description of no smoking |
| coll | Otherwise, unknown |
| alli | |
| KO1 | |
| ġ. | |
| .1800 | |
| 1 St | |
| Š, | |
| A | |
| A of Lakeda. For hour of | |

### 5. **GENERAL STUDY CONSIDERATIONS**

#### 5.1. Descriptive statistics

For categorical and quantitative data, descriptive statistics shown in Table, 5.-1 and will be calculated.

Table (5) -1 Descriptive statistics to be calculated

| Data type | Summary Type | Statistics to be calculated |
|---|---|---|
| Categorical data | Frequency table | Number and percentage of patients |
| Quantitative data | Summary statistics | Number of patients, arithmetic mean, standard deviation, Minimum, 14 quantiles, median, 34 quantiles, maximum |
| 5.2. Display of nume Descriptive statistics a | rical values<br>re presented in a table forn | nat 5 -2 according to. |
| | Table: | s 5 -2 and Presentation of descriptive statistics |

#### 5.2. Display of numerical values

Tables 5 -2 and Presentation of descriptive statistics

| Descriptive statistics | Labeling | EIID, |
|---|---|---|
| Number of patients | Display as an integer. | |
| Percentage | Round to one decimal place. | (a) |
| Arithmetic mean, standard deviation quantiles, median, 34 quantiles | on, 14 minutes Round up to +2 significant digi | ts of data and present with +1 significant digits of data. |
| Min, Max | Display the data with the same nu | mber of significant digits as the data. |
| Hazard ratio, confidence interval o | f hazard ratio Round off to one decimal place. | |
| Interval | Cl | |

#### 5.3. Software Used for Aggregate Analysis

SAS ® System Release 9.4 Use the above.

#### 5.4. Significance level and confidence interval

Unless otherwise specified, the significance level for hypothesis testing will be two-sided 5% and the confidence interval will be two-sided 95%.

### 5.5. Handling of missing data

Categories of "Unknown/Not specified" should be added as needed.

### Handling of Outliers

Outliers will not be handled in a special way in principle.

### 6. **Analysis Methods**

#### 6.1. Patient composition

Patients excluded from study population
Number of patients in exposure and control groups
Analysis procedure: For the above analytical variables, frequencies will be tabulated. The number of patients included and excluded will be tabulated for each reason for inclusion and exclusion.

A Calculation of frequencies

62 Patient characteristics

Analysis population: Analysis population
Analysis item: 4.5 Covariates items

Age (years) (category) 1)

0-14, 15-24, 25-34, 35-44, 45-44

Age (years) (category) 2)

Age (years) (category) 3)

Analysis procedure: For the above analytical variables, frequency tabulation of categorical data and quantitative data

Summary statistics of data will be calculated. At that time, the standardized difference between groups was calculated for each item.

Yes

### 6.3. **Primary Analysis**

Analysis Analysis Sets

population: Outcome (definition) 2)

Outcome:

Follow-up period Period covered:

**Analysis Conventions:** The incidence of outcomes per 10,000 person-years was calculated for each exposure and control group.

Also, a Cox proportional hazards model will be used to calculate the hazard ratio with 95% confidence interval

referring to the control group.

Kaplan-Meier curve

Analysis Sets

population: Outcome (definition) 2)

Outcome:

Period covered: Follow-up period

Cumulative Incidence of Outcomes by Exposure and Control Group, Kaplan-Meier, and Plot curves. N **Analysis Conventions:** 

The number of risk groups, the number of outcomes, and the number of censored subjects will be calculated by exposure and control group.

(a)

### 2) SSRI and other risks

Analysis Analysis Set (Control Group)
population: Outcome (Definition) 2)

Outcome:

Period covered: Follow-up
Stratification
factors: SSRI

Escitalopram Oxalate

Sertraline Hydrochloride
Paroxetine Hydrochloride
Fluvoxamine Maleate

• Above, 2, and Use of more

than one type

Analysis Conventions: Incidence of outcome by stratification factor Estimate (/ 10,000 person-years)

3) Outcome (definition) 3)

Analysis Analysis Sets

population: Outcome (definition) 3)

Outcome:

Period covered: Follow-up period

Analysis Conventions: The incidence of outcomes per 10,000 person-years was calculated for each exposure and control group.

Also, a Cox proportional hazards model will be used to calculate the hazard ratio with 95% confidence interval

referring to the control group.

### 4) SSRI, different risk (definition), 3)

Analysis Set (Control Group)
population: Outcome (Definition) 3)

Outcome:

Period covered: Follow-up
Stratification
factors: SSRI

· Escitalopram Oxalate

Sertraline Hydrochloride

· Paroxetine Hydrochloride

· Fluvoxamine Maleate

· Above, 2, and Use of more than one type

Analysis Conventions: Incidence of outcome by stratification factor Estimate (/ 10,000 person-years)

### 6.5. Sensitivity analyses

The same analysis as the primary analysis will be performed with the following conditions.

1) Change of the look back period and Change of

After changing the look back period to 1 year and (days) from the day before the Index Date to the past 1 year and (360 days), the analysis set (analysis set [sensitivity analysis 1]) will be reorganized, and the same analyses as the figure of patient composition, patient background, and primary analysis will be performed.

Changes in Gap Period and Grace Period and

After changing the Gap Period and Grace Period to up to 90 days, the analysis set (analysis set [sensitivity analysis 2)) will be reorganized, and the same analyses as the figure of patient composition, patient background, and primary analysis will be performed.

#### 3) Change in outcome definition

The same analysis as the primary analysis will be performed for the outcome (definition 1) and outcome (modified definition 2\*).

\*Definition, 2 and were changed to (1) to (3) below.

- (1) The definition of the same hospitalization is "the same 'Receipt ID or hospitalization in the month following the start of hospitalization 'Receipt ID."
  - (2) For drugs, only injections are applicable.
  - 3 Suspect flag is not considered for injuries/diseases

#### 4) Adjustments for propensity score

Analyzed:

Outcome: Outcome (definition) 2)

Period covered:

Analysis Conventions:

variables

Follow-up period
Logistic regression with the cohort as an objective variable, COV 1~3 and covariates of COV as explanatory

The propensity score will be estimated for each patient using the model, and the hazard ratio for the control group will be calculated using the Cox proportional hazards model with the for propensity score in the model. proparty of Takeda. For non-commercial use only and subject to

### 7. APPENDICES

#### 7.1. References

- 1) Christel R, et al., Association of Selective Serotonin Reuptake Inhibitors With the Risk for Spontaneous IntracranialHemorrhage. JAMA

- JAMA

  Sample Size Design for Medicine Kyoto University Academic Press

  4) Sacco R, et al. An updated definition of stroke for the 21st Century. A statement for healthcare professionals from the American Heart Association/American Stroke Association. Strok Epi 2013; 44: 2064 -2089.

  5) Kazuya F, et al., Accuracy of Japanese claims data in identifying diabetes-related complication. Stroke Association of Stroke Association. Stroke Association data in identifying diabetes-related complication.

- Property of Takeda. For noncommercial use only and subject to the applications of the property of takeda. 7) Masao I, et al., Gastrointestinal bleeding risk of selective serotonin reuptake inhibitors by level of kidney function: A population-based cohort study. Br

17/18

### 7.2. Induction rules, statistical methods

Tables 7 -1 and Analytical Handling

| Item | Definition |
|---|---|
| Look back period | From Day – 180 to 1 Day Before Index Date |
| | Injuries and illnesses are judged "on a monthly basis." |
| | Specifically, the 6 months before the month to which the Index Date belongs - the month to which the Index Date belongs - will be considered as the target period. |
| | in s |
| Look back period (sensitivity analysis 1 | L): Period from day – 360 to the day before the index date |
| | Injuries and illnesses are judged "on a monthly basis." |
| | Specifically, the target period is determined to be the month to which the Index Date belongs, which is 12 months before the month to which the Index Date belongs. |
| | Yes. |
| Duration of prescription | Prescription continuation period is the period from the day after the Index Date to 30 days after the final prescription |
| completion date (grace period). | |
| | Yes. If the interval (gap period) between consecutive prescription periods is $\leq 30$ days, it will be considered as |
| | prescription continued. If the interval (gap period) between consecutive prescription periods is $\geq 31$ days, it will be |
| Age calculated in the following manner. | The first day of the month of birth of an enrollee will be considered as the birth date, and the age on the Index Date will be |
| calculated in the following manner. | |
| | 350 |
| | ■Index if the birth date of the year has passed (Date of birth (month and day), Index date Date of birth (month and day)) |
| | Index date, Year of year of 1 year of birth |
| | ■Index If the birth date in the year has not passed (month and day of birth) > Index date month and day of |
| | Index Date Year of – Year of Birth Date -1 |
| Incidence rate (/ 10 ( | 2000 patient-years) = (Number of patients/Total follow-up period of target patients) X10000 * The total follow-up period of target |
| Incidence (person-year method) | patients should be summed up by the number of days and then divided by 365.25. |
| | Me and the second secon |
| < | O' |
| , 01 | |
| <b>~</b> 0 | |
| À. | |
| e O.C | |
| Ke | |
| 7.0 | |
| 7 | |
| dof Takedai. For S | |